CLINICAL TRIAL: NCT06536764
Title: Effects of Progressive Muscle Relaxation Exercises on Lumbopelvic Pain and Insomnia During Pregnancy.
Brief Title: Effects of Progressive Muscle Relaxation Exercises During Pregnancy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ayesha Razzaq
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Lumbopelvic Pain; Insomnia
Keywords: Lumbopelvic pain; Insomnia; Pregnancy; Progressive Muscle Relaxation Exercises
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: There will be comparison between two groups, experimental and control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): This group will receive Conventional therapy (hot pack, TENS, patient education) & Progressive muscle Relaxation exercises on low back 2 sessions per week for 6 weeks.
  Interventions: Other: Progressive Muscle Relaxation Exercises
- Control Group (Active Comparator): This group will receive Conventional therapy 2 sessions per week for 6 weeks. Conventional therapy involves hot pack, TENS and patient education.
  Interventions: Other: Conventional Therapy(Hot pack,TENS,Patient Education)

INTERVENTIONS:
Other: Progressive Muscle Relaxation Exercises — Progressive muscle Relaxation exercises will be performed by this group.Advise women to sit in chair. The therapist's voice will then instruct them to contract and release different muscle groups. They will practice tensing a muscle group until they feel the slight contraction and then release it, simultaneously contracting and relaxing all other muscle groups.Practice will progress in the same manner, starting with the muscles in the feet, then the calf, thigh, gluteal muscles, abdomen, chest, hands, forearms, arms, shoulders, neck, face, and finally the forehead muscles .
  Arms: Interventional group
Other: Conventional Therapy(Hot pack,TENS,Patient Education) — Conventional therapy including hot pack and TENS will be applied for 10 minutes each. Meanwhile, patients will be given education to ease back pain and improve sleep.
  Arms: Control Group

SUMMARY:
Lumbopelvic pain (LPP) during pregnancy is defined as pregnancy-related low back, or pelvic girdle pain. Pregnancy is a significant time for sleep disruptions as well.PMR involves systematically tensing and relaxing different muscle groups in the body, starting from the feet or hands and progressing through the body. This study aims to evaluate the impact of progressive muscle relaxation (PMR) exercises on the alleviation of low back pain and sleeplessness in pregnant women in their pregnancy.

DETAILED DESCRIPTION:
Literature suggests that Pregnancy involves hormonal and biomechanics adjustments, leading to changes in body systems for a secure fetus development. Painful symptoms and sleep disorders are common complaints, often present in the same individual.The exact cause of low back pain during pregnancy is not fully understood, but it is often linked to biomechanical, vascular, and hormonal changes.In the third trimester, 98% of women experience sleep difficulties, primarily caused by backache, urinary frequency, fetal movements, GERD, and leg discomfort.

The PMR technique involves deep breathing and progressive relaxation (tense-release) of major muscle groups. The technique promotes systematic relaxation of the major muscle groups of the body with the goal of physical and mental relaxation, reducing the response to stress, reducing skeletal muscle contractions, and decreasing pain sensations.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females with Age 20-40 years.During second and third trimester with
* Uncomplicated pregnancies.Pregnancy related LBP >3 on NPRS & Insomnia severity index (ISI) >10 score.Posterior lumbopelvic pain

Exclusion Criteria:

* Patients with Anterior Lumbopelvic Pain.
* Hemodynamically significant heart disease,
* Restrictive lung disease,
* Incompetent cervix/cerclage,
* Multiple gestation at risk for premature labor & Persistent bleeding.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Changes from Baseline to 6 weeks
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Pittsburgh Sleep Quality Index (PSQI) | Changes from Baseline to 6 weeks.
  The PSQI has 19 self-rated questions and five questions rated by a roommate or bed partner. The self-rated questions are combined into seven component scores, each with a range of 0-3, with 3 indicating the greatest dysfunction. The component scores are then added together to produce a global score, with a range of 0-21 points, with 0 indicating no difficulty and 21 indicating severe difficulties in all areas. Higher scores indicate worse sleep quality.
Insomnia severity index | Changes from Baseline to 6 weeks
  The questionnaire uses Likert -type scales to rate each element, with scores ranging from 0 to 4, with higher scores indicating more severe insomnia symptoms.Total score of 0-7 indicating no significant insomnia, 8-14 indicating sub threshold insomnia, 15-21 indicating clinical insomnia (moderate severity), and 22-28 indicating clinical insomnia (severe).

SECONDARY OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire | Changes from Baseline to 6 weeks
  This tool is used to assess the functional status of patients with low back pain, assessing ten daily functions and scoring them on a 0-5 scale, with the highest scoring statement indicating the true disability.0 - 4 indicationg No disability,5 - 14 Mild disability,15 - 24 Moderate disability ,25 - 34 Severe disability and 35 - 50 means Completely disabled.
Short Form-36 | Changes from Baseline to 6 weeks
  The questionnaire consists of 36 items assigned to 8 subscales.These 8 scales are further clustered into the physical component summary (physical function, role physical, bodily pain, and general health) and the mental component summary (vitality, social function, role-emotional, and mental health).High scores on all subscales indicate deterioration in QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PhD, Study Chair — Ripha International University, Islambad, Pakistan; Ayesha Razzaq, MSPT, Principal Investigator — Ripha International University, Islambad, Pakistan
Locations (1):
- Samra Yosaf Materniy Clinic, Mirpur, Azad Jammu & Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No